CLINICAL TRIAL: NCT05567328
Title: Validation of the New Vibration-guided FibroScan Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M140
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Liver Diseases
Keywords: FibroScan; Vibration Control Transient Elastography; Vibration Guided Transient Elastography; Liver Stiffness Measurement; VCTE; VGTE
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patient (age >= 18 y.o) followed for a liver disease, all etiologies combined (Experimental): Adult patients followed in the Hepatology or Endocrinology department for a liver disease, all etiologies combined.
  Interventions: Device: Research FibroScan (FS)

INTERVENTIONS:
Device: Research FibroScan (FS) — Exams will be performed with the M or XL probe as per FS recommendations. Same probe must be used for all exams Exploratory exam after patient 151 are performed with adapted view of Research FS
  Patients 1 to 90 & 151 to 190 Exam1 Exploratory exam with the Research FS Exam2 Reference exam with the CE-marked FS
  Patients 91 to 130 & 191 to 230 Exams1&2 Two consecutive Exploratory exams with the Research FS Exams3&4 Two consecutive Reference exams with the CE-marked FS
  Patients 131 to 150 Exams1&2 Two consecutive Exploratory exams with automatic function of the Research FS Exam3 Reference exam with the CE-marked FS
  Patients 231 to 270 Exams1 (novice operator) Exploratory exam with the Research FS Exams2 (novice operator) Reference exam with the CE-marked FS Exams3 (experienced/expert operator) Exploratory exam with the Research FS Exams4 (experienced/expert operator) Reference exam with the CE-marked FS

SUMMARY:
This is an European, prospective, interventional, multicenter clinical investigation that will take place in 2 French sites. 100 adults patients will be included. The study objective is to compare the applicability between the Research FibroScan and the reference FibroScan examination performed on the liver.

DETAILED DESCRIPTION:
Chronic liver disease (CLD) is a silent disease that can progress to life-threatening conditions. Hepatitis B (HBV) and C (HCV) viruses, alcoholic liver disease (ALD) and non-alcoholic fatty liver disease (NAFLD) are the main causes of chronic liver inflammation.

CLDs represent a major public health burden, with global estimates showing around a rate of 2 million deaths per year, including 1 million from complications of cirrhosis and 1 million from viral hepatitis and hepatocellular carcinoma. About 75 million people are diagnosed with alcohol use disorders and are at risk of developing alcohol-related liver disease. About 2 billion adults are obese or overweight and more than 400 million suffer from diabetes; both of which are risk factors for the development of NAFLD and HCC.

NAFLD is currently the leading cause of CLD worldwide with a reported worldwide prevalence of 25% in adults. Early identification among NAFLD patients with non-alcoholic steatohepatatis (NASH) and advanced fibrosis is particularly important as they are at high risk of developing liver complications. The main difficulty in diagnosing NASH patients is related to their symptomatology, which is not always clinically useful because it is not specific. Therefore a screening for advanced stage of NAFLD is recommended in patient at high risk such patients with type 2 diabetes or obesity.

Liver fibrosis is known to be a major prognostic predictor of hepatic and overall mortality in patients with CLD. Therefore, early diagnosis of liver fibrosis is crucial in asymptomatic individuals.

Liver biopsy (LB) is the gold standard diagnostic test for the evaluation of patients with CLD. However, it is difficult to use it as a screening tool given the large number of patients with NAFLD.

The development of non-invasive and broadly applicable screening tools for the assessment of liver fibrosis appears to be a major public health opportunity.

Among the non-invasive tools available, the FibroScan (Echosens™, Paris, France) has proven to be a useful tool for diagnosing fibrosis and steatosis in patients with CLD. FibroScan is a device based on Vibration-Controlled Transient Elastography (VCTE™) technology that measures Liver Stiffness Elasticity (LSM) to assess fibrosis and Controlled Attenuation Parameter (CAP) to assess steatosis.

In this context, Echosens aims to develop a new technology called "Vibration-Guided Transient Elastography (VGTE)" which is an original method that will help FibroScan operators to localize an optimal region of interest for stiffness measurement in a simple and reliable way.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > = 18 years old) followed for a liver disease; a suspicion of liver disease or for consequences of liver disease, all etiologies combined
* Patient must be able to give written informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Vulnerable patient
* Patients with ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Difference of patient percentage having a successful examination between the novel and the reference FibroScan examination | 17 months
  To compare the applicability between the novel FibroScan and the reference FibroScan examination performed on the liver

SECONDARY OUTCOMES:
Difference of success rate between the novel and the reference FibroScan examination | 17 months
  To compare the success rate between the novel and the reference FibroScan examination
Difference between the initial localization durations required for the novel and the reference FibroScan examination. | 17 months
  To compare, between the novel and the reference examination, the duration of the initial localization, defined between the time the operator places the probe on the patient and the time needed to obtain the first valid stiffness measurement
Difference between the examination durations required for the novel and the reference examination based on liver stiffness measurements. | 17 months
  To compare between the novel and the reference examination the duration between the time of the operator places the probe on the patient and the time he obtains 10 valid liver stiffness measurements
Difference between the examination durations required for the novel and the reference examination based on CAP measurements. | 17 months
  To compare between the novel and the reference examination, the duration between the time of the operator places the probe on the patient and the time he obtains the CAP value with the gauge at 100%.
Intraclass Correlation Coefficient (ICC) between novel and reference FibroScan examinations | 17 months
  To compare the agreement of CAP, stiffness and skin to capsule distance (SCD) between the novel and the reference examination
Evaluation of the operator perception between the novel and reference examination | 17 months
  To compare with a dedicated questionnaire (quantitative scale), the operator perception related to the probe vibration, indicator display and easy of use.
Evaluation of the patient perception between the novel and reference examination | 17 months
  To compare with a dedicated questionnaire (quantitative scale), the patient perception related to the probe vibration
ICC between the two novel FibroScan examinations and the two reference FibroScan examinations and coefficient of repeatability of stiffness and CAP examination performed by the same operator, on the same patient the same day. | 17 months
  To evaluate the repeatability (same day, same operator) of the stiffness and the CAP measurements of the novel and the reference examinations
ICC between novel and reference FibroScan examinations based on the operator's level expertise and coefficient of reproducibility of stiffness and CAP examination performed by the 2 different operators, on the same patient the same day. | 17 months
  To evaluate the inter-operator reproducibility of the stiffness and the CAP measurements of the novel and the reference examination, based on the operator's level of expertise.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Beaujon, Clichy
  - Hospices Civils de Lyon - Lyon Sud, Lyon
  - CHU de Nancy, Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bastard C, Audiere S, Foucquier J, Loree H, Miette V, Bronowicki JP, Stern C, Caussy C, Sandrin L. Guided-VCTE: An Enhanced FibroScan Examination With Improved Guidance and Applicability. Ultrasound Med Biol. 2025 Apr;51(4):628-637. doi: 10.1016/j.ultrasmedbio.2024.12.007. Epub 2025 Jan 13. PMID 39809636